CLINICAL TRIAL: NCT05173584
Title: Is Levalbuterol an Effective Treatment With Less Cardiac Side Effects Than Albuterol in Hyperkalemia Patients: A Randomized-controlled Clinical Trial Protocol.
Brief Title: Levalbuterol Compared to Albuterol Regarding Cardiac Side Effects and Potassium Lowering Effects.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aleppo (Other)
Responsible Party: Principal Investigator, Baraa Shebli, Cardiology Resident, University of Aleppo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15993
Record Dates: First submitted 2021-11-24; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Hyperkalemia
Keywords: Hyperkalemia; Albuterol; Levalbuterol; Heart rate
MeSH Terms: conditions — Hyperkalemia | interventions — Levalbuterol; Albuterol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levalbuterol Arm (Experimental)
  Interventions: Drug: Levalbuterol
- Albuterol Arm (Active Comparator)
  Interventions: Drug: Albuterol

INTERVENTIONS:
Drug: Levalbuterol — Levalbuterol nebulizer solution 1.25mg/3ml with a total dose of 5 mg (12ml) for each patient.
  Arms: Levalbuterol Arm
Drug: Albuterol — Albuterol nebulizer solution 2.5 mg/3ml with a total dose of 0 mg (12ml) for each patient.
  Other Names: salbutamol, racemic albuterol
  Arms: Albuterol Arm

SUMMARY:
Hyperkalemia is a common life-threatening electrolyte disturbance which may impair cardiac and many other organs' functions. Unfortunately, a well-established guideline for the treatment of hyperkalemia in the emergency setting is still missing. However, the last "Kidney Disease: Improving Global Outcomes (KDIGO)" conference proposed a treatment protocol for hyperkalemia and addressed controversies in this matter. Beta2-agonists were one of the main lines in the approach towards managing a patient with hyperkalemia. However, this evidence was only available for racemic albuterol.

Levalbuterol is the isolated R-enantiomer of racemic albuterol which is comprised of S- and R-enantiomers. Several lab and clinical studies have assessed the effect, affinity, and selectivity of each of the enantiomers. Few studies in medical literature have compared the difference between these two drugs regarding cardiac effects with inconclusive results, and even fewer studies have compared the efficacies of these two drugs regarding potassium lowering effect.

To the investigators' knowledge, no study to date has compared the efficacy and safety of albuterol compared to levalbuterol in hyperkalemic patients with the properly adjusted dosing. So, in clinical practice, the investigators wanted to know based on evidence if levalbuterol can be an effective substitute for albuterol in lowering potassium levels in hyperkalemia patients while yielding fewer cardiac side effects. To answer this question, the investigators designed a single-centered controlled clinical trial that includes adult hyperkalemia patients in Aleppo University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* serum potassium level >5.9 mEq/L

Exclusion Criteria:

* Pseudohyperkalemia:

  * Hemolysis of blood sample
  * Thrombocytosis > 10*6 /mm3
  * Hyperleukocytosis > 10*5/mm3
  * Mechanical Trauma during Venipuncture
  * Fist clenching during blood drawing
  * Tourniquet time > 1 minute
* Diabetes acute complications

  * DKA
  * Hyperosmolar Hyperglycemic Syndrome
* Insulin-dependent diabetes mellitus ( if insulin is taken recently)
* Pregnant women
* Hyperthyroidism
* Hemodynamic instability
* Pacemakers if providing impulses (demand pacemakers that are not firing right now are included)
* Atrial fibrillation or any other arrhythmia
* Baseline tachycardia >120 bpm
* Acute exacerbations of HF
* Patients expected to require emergency intubation and ventilation
* Patients expected to require dialysis within the first 60 minutes
* Patients with hypersensitivity to the medication
* Patients with Acute Coronary Syndrome
* Patients on beta-blockers / beta-agonists or anti-arrhythmic drugs
* Patients with severe dyspnea or hypoxia SpO2 <90%

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate changes | Heart rate is measured at baseline before drug administration and at 15, 30, 45, 60, 90, 120 minutes after treatment.
  Heart rate changes over time measured as beats per minute
Serum potassium level changes | Serum potassium levels are measured at baseline and 90 minutes after treatment administration
  Serum potassium level changes after treatment measured as mEq/L

SECONDARY OUTCOMES:
ECG changes | ECG changes detected at baseline and at 90 minutes after therapy
  ECG Changes at presentation with hyperkalemia (Depressed ST segment, Diphasic T wave, Prominent U wave, Peaked T wave, Wide PR interval, Wide QRS duration, Peaked T wave, Loss of P wave, Sinusoidal wave, Others) and after treatment
Blood Pressure (BP) changes | BP changes measured at baseline and at 30, 60, and 90 minutes after therapy
  BP changes over time measured as mmHg
Frequency of reported symptoms at presentation | Symptoms reported only at the presentation of the patient
  Symptoms at presentation (Muscle weakness, Paresthesia, Paralysis, flushing, Nausea/Vomiting, Chest pain, Dyspnea, Fasciculation, Palpitations, Others).
Frequency of Adverse effects | Adverse effects after treatment detected during the first two hours following treatment
  Adverse effects following treatment (Fever, Palpitations, Hypoglycemia, Hypokalemia, Headache, Tremor, Nervousness, Nausea/vomiting, Lightheadedness)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Malhis, MRCP, Study Director — Professor of Cardiology, Head of Cardiology division, Aleppo University Hospital, Faculty of Medicine, University of Aleppo.; Baraa Shebli, M.D., Principal Investigator — Cardiology Resident, Aleppo University Hospital, Faculty of Medicine, University of Aleppo
Locations (1):
- Aleppo University Hospital, Aleppo, Aleppo Provice, Syria

REFERENCES:
- [Derived] Shebli B, Ghabally M, Shabouk MB, Arnaout AY, Zeina MB, Malhis M. Assessing the cardiovascular and potassium lowering effects of levalbuterol compared to albuterol: a randomized control trial. Front Cardiovasc Med. 2025 Dec 8;12:1463999. doi: 10.3389/fcvm.2025.1463999. eCollection 2025. PMID 41437987